CLINICAL TRIAL: NCT01774981
Title: Study of the Safety and Efficacy of LY3016859 After Multiple Intravenous Dosing in Diabetic Nephropathy Patients
Brief Title: Study of LY3016859 in Participants With Diabetic Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14353; I5V-MC-TGAB (Other: Eli Lilly and Company); 2012-004496-40 (EudraCT Number)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo (Part A) (Placebo Comparator): Part A: Placebo administered by 60 minute Intravenous (IV) infusion at Week 1 and Week 4.
  Interventions: Drug: Placebo
- 10 mg LY3016859 (Part A) (Experimental): Part A: 10 milligram (mg) LY3016859 administered by 60 minute IV infusion at Week 1 and Week 4.
  Interventions: Drug: LY3016859
- 100 mg LY3016859 (Part A) (Experimental): Part A: 100 mg LY3016859 administered by 60 minute IV infusion at Week 1 and Week 4.
  Interventions: Drug: LY3016859
- 750 mg LY3016859 (Part A) (Experimental): Part A: 750 mg LY3016859 administered by 60 minute IV infusion at Week 1 and Week 4.
  Interventions: Drug: LY3016859
- Placebo (Part B) (Placebo Comparator): Part B: Placebo administered by 60 minute IV infusion at Weeks 1, 4, 7, 10 and 13.
  Interventions: Drug: Placebo
- 50 mg LY3016859 (Part B) (Experimental): Part B: 50 mg LY3016859 administered by 60 minute IV infusion at Weeks 1, 4, 7, 10 and 13.
  Interventions: Drug: LY3016859
- 250 mg LY3016859 (Part B) (Experimental): Part B: 250 mg LY3016859 administered by 60 minute IV infusion at Weeks 1, 4, 7, 10 and 13.
  Interventions: Drug: LY3016859
- 750 mg LY3016859 (Part B) (Experimental): Part B: 750 mg LY3016859 administered by 60 minute IV infusion at Weeks 1, 4, 7, 10 and 13.
  Interventions: Drug: LY3016859

INTERVENTIONS:
Drug: Placebo — Administered IV
  Arms: Placebo (Part A); Placebo (Part B)
Drug: LY3016859 — Administered IV
  Arms: 10 mg LY3016859 (Part A); 100 mg LY3016859 (Part A); 250 mg LY3016859 (Part B); 50 mg LY3016859 (Part B); 750 mg LY3016859 (Part A); 750 mg LY3016859 (Part B)

SUMMARY:
The purpose of this two-part study is to investigate the safety, tolerability and efficacy of LY3016859 after multiple intravenous (IV) dosing's in participants with diabetic nephropathy (DN). Part A will be dose escalation for safety and tolerability and Part B will evaluate Proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Stable diabetic kidney disease (DKD) while taking Standard of Care medication (SOC), as defined by:

  * Estimated glomerular filtration rate (eGFR) less than (<) 90 milliliter per minute per 1.73 square meter (ml/min/1.73m²) as determine utilizing the Modification of Diet in Renal Disease (MDRD) equation
  * Taking an angiotensin convertible enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB) at a stable dose for greater than or equal to (≥) 2 months prior to randomization and agree to continue to take such throughout the duration of the study
  * Type 1 or Type 2 diabetes on a stable treatment regimen and adequately controlled in the opinion of the investigator
  * First morning protein-creatine ratio (PCR) at screening ≥400 milligrams per gram (mg/g) (Part B only)
* Clinical chemistry labs within acceptable range for the participant population, as per investigator judgment
* Men and women of non-childbearing potential as determined by medical history and physical examination

  * Non-vasectomized male participants must agree to use a medically accepted method of contraception with all sexual partners during the study and for 90 days following the final dosing. Medically accepted effective forms of contraception may include condoms with contraceptive foam or having partners use diaphragms with contraceptive jelly or cervical caps with contraceptive jelly
  * Female participants must be postmenopausal or surgically sterile to participate in this study. This is defined as females between age 45 to 75 years, inclusive, and either 12 months without a menstrual period [no follicle stimulating hormone (FSH) test required] or 6-12 months without a menstrual period and follicle stimulating hormone (FSH) greater than (>) 40 international units per liter (IU/L)
* Must weigh ≥50 kilograms (kg) at time of screening and dosing
* Acceptable sitting blood pressure (BP) per the following American Heart Association (AHA) guidelines:

  * Normal: systolic blood pressure (SBP) <120 millimeters of mercury (mmHg) and diastolic blood pressure (DBP) <80 mmHg
  * Prehypertension: SBP 120-139 or DBP 80-89
  * High Blood Pressure (Hypertension) Stage 1: SBP 140-159 mmHg or DBP 90-99
* Have given written informed consent prior to any study-specific procedures
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow site specific study procedures
* Have venous access sufficient to allow blood sampling
* Have laboratory values and other safety parameters that are, in the opinion of the investigator, acceptable fo participation for the study

Exclusion Criteria:

* Have a diagnosis of chronic kidney disease (CKD) other than DKD, (hypertensive nephrosclerosis superimposed on DKD is acceptable)
* Have SBP >160 mmHg or DBP >100 mmHg

  o Individuals with Stage 1 BP elevation (SBP 140-159 mmHg or DBP 90-99 mmHg) on some occasions during study, may be acceptable, as long as only non-protein-lowering antihypertensives are adjusted to achieve target BP goals (<140/90 mmHg)
* Current use of (or within 2 weeks of enrollment), or projected need for a renin inhibitor or aldosterone antagonist, or a combination of Angiotensin-converting enzyme inhibitors/angiotensin II receptor blockers (ACEi/ARB)
* Individuals in whom dialysis or transplantation is anticipated within 6 months of screening
* Have a history of acute kidney injury within 3 months of screening
* Are currently enrolled in, or discontinued within the last 60 days from, a clinical trial involving an investigational drug that has not received regulatory approval for any indication and/or have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives of the administered drug (whichever is longer) prior to dosing
* Have previously completed or withdrawn from this study or any other study investigating LY3016859
* Have a diagnosis of Class III or IV congestive heart failure (as defined by the New York Heart Association)
* Have an abnormality in the 12-lead Electrocardiogram (ECG) that, in the opinion of the investigator increases the risks associated with participating in the study. In addition, individuals with the following findings will be excluded:

  * Confirmed corrected QT (QTcF) interval >450 milliseconds (msec) for men and >470 msec for women
  * Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular ectopic beats
  * History of unexplained syncope
  * Family history of unexplained sudden death or sudden death due to long QT syndrome
  * T-wave configurations are not of sufficient quality for assessing QT interval, as determined by the investigator
* Have evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies; have a history of cirrhosis or hepatitis C or are positive for hepatitis C antibody at the screening visit; are known to be hepatitis B surface antigen-positive or are positive for hepatitis B surface antigen at the screening visit
* Are unwilling to discontinue use of Chinese herbs for at least 2 weeks prior to randomization and for the duration of their study participation
* Are unwilling or unable to comply with the use of a data collection device to directly record data from the participant
* Have donated blood of more than 500 milliliters (mL) within the last 60 days prior to screening
* Have an average weekly alcohol intake that exceeds 21 units per week or are unwilling to stop alcohol intake within 48 hours of entry into study and for the duration of the study (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Individuals who, in the opinion of the investigator, show evidence of regular use of drugs of abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLilly (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST_, Study Director — Eli Lilly and Company
Locations (7):
- United States (6):
  - Innovative Research of West Florida, Clearwater, Florida
  - Creighton University Medical Center, Omaha, Nebraska
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - TAD Clinical Research, Lufkin, Texas
  - Renal Associates, PA, San Antonio, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo (Part A) | 10 mg LY3016859 (Part A) | 100 mg LY3016859 (Part A) | 750 mg LY3016859 (Part A) | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B)
Started | 3 | 4 | 4 | 4 | 6 | 14 | 13 | 12
Received at Least 1 Dose of Study Drug | 3 | 4 | 4 | 4 | 6 | 14 | 13 | 12
Completed | 3 | 4 | 4 | 4 | 5 | 13 | 13 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 100 mg LY3016859 (Part A): Part A:100 mg LY3016859 administered by 60 minute IV infusion at Week 1 and Week 4.
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | 10 mg LY3016859 (Part A) | 100 mg LY3016859 (Part A) | 750 mg LY3016859 (Part A) | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B) | Total
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 6 | 14 | 13 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10.0) | 57 (7.2) | 56 (6.1) | 62 (11.6) | 55 (5.0) | 63 (8.3) | 55 (12.7) | 59 (9.5) | 58.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 5 | 7 | 4 | 6 | 28
  Male | 2 | 3 | 2 | 2 | 1 | 7 | 9 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 5 | 10
  Not Hispanic or Latino | 3 | 4 | 4 | 4 | 5 | 10 | 13 | 7 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  White | 3 | 4 | 4 | 4 | 6 | 12 | 13 | 12 | 58
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 2 | 0 | 0 | 3 | 10 | 13 | 9 | 37
  Bulgaria | 1 | 2 | 3 | 2 | 3 | 4 | 0 | 3 | 18
  United Kingdom | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part B:Change From Baseline in Proteinuria
Description: Proteinuria is defined as the ratio of protein to creatinine.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who received at least one dose of study drug in Part B with a baseline measurement and at least one post-baseline measurement.
Measure: Mean (Standard Deviation); unit: grams per 12 hour (g/12 hour)
Arm/Group | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B)
Number analyzed (Participants) | 6 | 9 | 9 | 11
grams per 12 hour (g/12 hour) | 1.5 (2.04) | -0.4 (1.60) | 0.1 (1.21) | 0.7 (2.23)
Statistical Analysis 1: Comparison: Placebo (Part B) vs 50 mg LY3016859 (Part B); Test type: Superiority or Other; p = 0.0449, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo (Part B) vs 250 mg LY3016859 (Part B); Test type: Superiority or Other; p = 0.0808, t-test, 1 sided
Statistical Analysis 3: Comparison: Placebo (Part B) vs 750 mg LY3016859 (Part B); Test type: Superiority or Other; p = 0.2219, t-test, 1 sided

2. Primary Outcome: Part A and Part B: Number of Participants With One or More Treatment Emergent Adverse Events (AEs) or Any Serious AEs
Description: Treatment-emergent adverse events (TEAEs) are events which were not present at baseline or pre-existing conditions at baseline that worsened in severity following the start of treatment. A summary of other non-serious Adverse Events (AEs), and all Serious Adverse Events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to 32 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg LY3016859 (Part A): Part A:10 milligram (mg) LY3016859 administered by 60 minute IV infusion at Week 1 and Week 4.
Arm/Group | Placebo (Part A) | 10 mg LY3016859 (Part A) | 100 mg LY3016859 (Part A) | 750 mg LY3016859 (Part A) | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B)
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 6 | 14 | 13 | 12
Participants | 1 | 3 | 4 | 2 | 6 | 13 | 13 | 11

3. Secondary Outcome: Part B: Change From Baseline in Proteinuria Over Time
Description: Proteinuria is defined as the ratio of protein to creatinine.
Time Frame: Baseline, 19 Weeks
Population: All randomized participants who received at least one dose of study drug and were in Part B with a baseline measurement and at least one post-baseline measurement.
Measure: Mean (Standard Deviation); unit: mg/dl of protein/ by mg/dl of creatinine
Arm/Group | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B)
Number analyzed (Participants) | 5 | 11 | 12 | 11
mg/dl of protein/ by mg/dl of creatinine | 19.3 (154.66) | -17.3 (81.95) | -2.4 (88.01) | 48.6 (130.13)

4. Secondary Outcome: Part B: Change From Baseline in Albuminuria Over Time
Description: Albuminuria is defined as the ratio of albumin to creatinine.
Time Frame: Baseline, 19 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dl of albumin/ by mg/dl of creatinine
Groups:
- Placebo (Part B): Part B:Placebo administered by 60 minute IV infusion at Weeks 1, 4, 7, 10 and 13.
Arm/Group | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B)
Number analyzed (Participants) | 5 | 11 | 12 | 11
mg/dl of albumin/ by mg/dl of creatinine | 8.6 (100.57) | -15.6 (64.27) | -8.1 (50.19) | 36.7 (93.49)

ADVERSE EVENTS:
Arm/Group | Placebo (Part A) | 10 mg LY3016859 (Part A) | 100 mg LY3016859 (Part A) | 750 mg LY3016859 (Part A) | Placebo (Part B) | 50 mg LY3016859 (Part B) | 250 mg LY3016859 (Part B) | 750 mg LY3016859 (Part B)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 0/4 | 1/6 | 0/14 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 0/4 | 1/6 | 3/14 | 6/13 | 2/12
Other Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 4/4 | 2/4 | 6/6 | 13/14 | 13/13 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=3) | 10 mg LY3016859 (Part A) (N=4) | 100 mg LY3016859 (Part A) (N=4) | 750 mg LY3016859 (Part A) (N=4) | Placebo (Part B) (N=6) | 50 mg LY3016859 (Part B) (N=14) | 250 mg LY3016859 (Part B) (N=13) | 750 mg LY3016859 (Part B) (N=12)
Anginal pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation aggravated (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phytobezoar (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acalculous cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic lower extremity cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoropopliteal artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=3) | 10 mg LY3016859 (Part A) (N=4) | 100 mg LY3016859 (Part A) (N=4) | 750 mg LY3016859 (Part A) (N=4) | Placebo (Part B) (N=6) | 50 mg LY3016859 (Part B) (N=14) | 250 mg LY3016859 (Part B) (N=13) | 750 mg LY3016859 (Part B) (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia aggravated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heart pounding (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cloudy vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tearing decreased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal fullness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Distress gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry heaves (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Application site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coldness general (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Edema generalized (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General body pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of legs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein phlebitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hay fever (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha hemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection due to unspecified staphylococcus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis of hand (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leg infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract yeast infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abrasions (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
First degree burns (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flea bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spider bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sprained ankle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bicarbonate decreased serum (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol levels raised (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecg abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fasting blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased intraocular pressure (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelets decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Potassium abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Uric acid level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appetite lost (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fasting hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout aggravated (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout flare (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia aggravated (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metabolic acidosis worsened (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volume depletion (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Volume overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain in thumb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Headache aggravated (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica aggravated (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression worsened (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Difficulty sleeping (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney function abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough nonproductive (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supine dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Localised rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Localized erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mohs micrographic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood pressure high (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing of face (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension exacerbated (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension worsened (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infusion Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crawling Sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Numbness in Feet (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days